CLINICAL TRIAL: NCT06075875
Title: Comparative Study Between Vegetable Proteins, and Mixed Animal Proteins on the Outcome of Hepatic Encephalopathy Patients in ICU and Wards
Brief Title: Vegetable Proteins Versus Mixed Animal Proteins on the Outcome of Hepatic Encephalopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Hepatology & Tropical Medicine Research Institute (Other Government)
Responsible Party: Principal Investigator, ICU, fellow of intensive care medicine, National Hepatology & Tropical Medicine Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 45-2023
Record Dates: First submitted 2023-08-29; First posted 2023-10-10 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Plant Proteins, Dietary

STUDY DESIGN:
Intervention Model Description: prospective, randomized, double blind,single-center study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control=mixed animal and vegetable proteins (Active Comparator): mixed animal and vegetable proteins in the standard ratio (2/3:1/3; 60%:40% respectively) present in the nutritional menu over all hospitals in the general organization of teaching hospitals and institutes "GOTHI"; Egypt= as a control group.(average 2000Kcal) and proteins 1.2g/Kg/day15 (average 84gm).
  Interventions: Dietary Supplement: mixed animal and vegetable proteins
- study= pure vegetable proteins (Experimental): pure vegetable proteins (a study group). (average 2000Kcal) and proteins 1.2g/Kg/day15 (average 84gm).
  Interventions: Dietary Supplement: pure vegetable proteins

INTERVENTIONS:
Dietary Supplement: mixed animal and vegetable proteins — mixed animal and vegetable proteins in the standard ratio (2/3:1/3; 60%:40% respectively) present in the nutritional menu over all hospitals in the general organization of teaching hospitals and institutes "GOTHI"; Egypt= as a control group) and continued for at least 48hours and followed for five days. The vegetable diets will be prepared from the dietetic service of our institute;calories will be calculated for 30Kcal/Kg/day (average 2000Kcal) and proteins 1.2g/Kg/day15 (average 84gm).
  Arms: control=mixed animal and vegetable proteins
Dietary Supplement: pure vegetable proteins — pure vegetable proteins continued for at least 48hours and followed for five days. The vegetable diets will be prepared from the dietetic service of our institute;calories will be calculated for 30Kcal/Kg/day (average 2000Kcal) and proteins 1.2g/Kg/day15 (average 84gm).
  Arms: study= pure vegetable proteins

SUMMARY:
Vegetables are thought to be beneficial not only because of their high content of fiber, which promotes bacterial fermentation and decreases colonic transit time, decreasing ammonia absorption from the gut, but also because of their high BCAA content, low methionine and tryptophan contents, and the induction of gut microbiota which, in turn, increases fecal nitrogen excretion. Also the fact supporting the underlying rationale for the use of vegetable proteins is that dietary fiber contributes to the improvement of glycemic control in these patients. Smaller sample studies also support the idea that vegetable based protein diets have better effect on cognition in patients with HE; in these studies vegetable protein diet was compared to meat protein diet and patients with HE showed improvement in cognition on former diets. However, no positive effects were shown by Shaw or Chiarino.

Similarly, another older single blind crossover study (n=10) showed that as compared to meat proteins, vegan diet has a better effect on mental status as determined on psychometric testing in patients with HE.

As a result of the limited studies and small number of participants of the effect of vegetable proteins on HE, the purpose of this study is to investigate the effects of a vegetable versus mixed animal and vegetable protein diet on hepatic encephalopathy.

DETAILED DESCRIPTION:
After approval by NHTMRI-IRB Ethical Committee.All demographic data will be obtained including the patients age, sex,associated co-morbidities (diabetes mellitus & hypertension), cause of hepatic encephalopathy, grade of hepatic encephalopathybythe West Haven criteria (WHC),14Child-Pugh score, Model for end stage liver disease (MELD) score, and subjective global assessment (SGA).

All patients will receive the routine medical supportive treatment of hepatic encephalopathy in the form of rectal enemas, oral non-absorbable disaccharides (Lactulose), non-absorbable antibacterial (Rifaximin).

All patients will receive enteral nutrition either oral if tolerated (HE grade I/II) or through nasogastric tubes (if intolerant; HE grade III/IV). Patients were assessed for 24 hours for tolerance of enteral feeding.

Patients were randomized to receiveeither diets containingpure vegetable proteins (a study group) versus the mixed animal and vegetable proteins in the standard ratio (2/3:1/3; 60%:40% respectively) present in the nutritional menu over all hospitals in the general organization of teaching hospitals and institutes "GOTHI"; Egypt= as a control group) and continued for at least 48hours and followed for five days. The vegetable diets will be prepared from the dietetic service of our institute;calories will be calculated for 30Kcal/Kg/day (average 2000Kcal) and proteins 1.2g/Kg/day15 (average 84gm).

Follow up daily for the degree of hepatic encephalopathy by WHC criteria will be recorded.Complete blood counts, urea, and blood glucose will be monitored in the first 72hours. Follow up arterial ammonia will e on day zero (start of regimen) and day three.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18years old
* admitted to the intensive care unit or wards of the National Hepatology and Tropical Medicine Research Institute (NHTMRI) who have or developed hepatic encephalopathy and have no contraindication for enteral nutrition

Exclusion Criteria:

* If they have contraindication for enteral nutrition e.g. intestinal obstruction, or active hematemesis.
* Patients who are on total parenteral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2023-12-23 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
grade of hepatic encepalopathy | 48hours
  if the vegetable proteins will improve the hepatic encephalopathy grade in comparison with animal proteins.

SECONDARY OUTCOMES:
length of stay | during the study up to 24 weeks
  ICU ength of stay
length of stay | during the study up to one year
  hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- NHTMRI, Cairo, Egypt